CLINICAL TRIAL: NCT06697964
Title: High Resolution Anuscopy Study
Status: Recruiting | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: HRA Study
Record Dates: First submitted 2024-09-19; First posted 2024-11-20 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Human Papilloma Virus; Anal Squamous Cell Carcinoma
MeSH Terms: conditions — Anus Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: HRA — High resolution anoscopy to help evaluate anal conditions such as precancerous lesions

SUMMARY:
The majority of anal squamous cell carcinomas (SCC) stem from infection with high-risk human papillomavirus (HPV). Anal SCC is rare among the general population but affects several populations disproportionately.

High-risk groups are screened through anal swabs for anal cytology and detection of high risk human papillomavirus (HR HPV). HRA referral is recommended for individuals with abnormal cytology.

HRA represents the only method to identify precancerous lesions of the anal canal, with only few specialists knowledgeable about it.

At UZ Brussel, the investigators collected a wealth of data about HPV infection and its association with anal pathology. By establishing a comprehensive study, the investigators can delve into this data with specific research questions, conducting valuable research to provide answers to pressing clinical questions and contribute to advancements in medical understanding and treatment.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have undergone HRA and all future patients referred for HRA in UZ Brussel
* 18 years or older
* Understands and able to speak and write in French, Dutch or English

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent or will undergo High Resolution Anoscopy in UZ Brussel after Informed Consent
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
comparison of the prevalence of precancerous lesions in men who have sex with men using PrEP or are HIV positive Men | Through study completion, on average 5 years
Exploration of associations between abnormal histology and patient characteristics | Through study completion, on average 5 years
comparison of the prevalence of precancerous lesions in different groups | Through study completion, on average 5 years
to delineate unique features associated with HSIL in each risk group by linking patterns or characteristics | Through study completion, on average 5 years
  such as verrucous aspects, coarse punctuation, mosaic patterns, flat morphology, and fragility
Prevalence of anal cancer among the at-risk populations | Through study completion, on average 5 years
correlation between abnormal histology and abnormal cytology, as well as HPV infection in MSM using PrEP and MSM living with HIV | Through study completion, on average 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Jette, Belgium

IPD SHARING:
Plan to Share IPD: No